CLINICAL TRIAL: NCT00861237
Title: Homeopathy for Prevention of Atrial Fibrillation After Aortocoronary Bypass Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Number of patients recruited to small, no cooperation of study members
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Frass, Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2342
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Atrial Fibrillation
Keywords: Nux vomica; homeopathy; heart lung machine; heart surgery; postoperatively studied
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo globules group (Placebo Comparator): Patients receive Placebo globules made out of sugar and looking similar to active drug sublingually before surgery.
  Interventions: Drug: Placebo (placebo comparator)
- Nux vomica group (Active Comparator): Patients receive Nux vomica globules made out of sugar sublingually before surgery.
  Interventions: Drug: Nux vomica (active comparator)

INTERVENTIONS:
Drug: Nux vomica (active comparator) — Patients receive Nux vomica in a homeopathic potentiation
  Other Names: Strychnos Nux vomica C200
  Arms: Nux vomica group
Drug: Placebo (placebo comparator) — Patients receive Placebo looking similar to active drug
  Other Names: Placebo globules
  Arms: Placebo globules group

SUMMARY:
After heart surgery, about 30% of patients suffer from atrial fibrillation. Patients are randomized into two groups receiving either potentized Strychnos Nux vomica or placebo under double blind conditions. Postoperatively, ECGs are done to monitor cardiac rhythm.

DETAILED DESCRIPTION:
Preoperatively, patients receive potentized Nux vomica or placebo sublingually. Then, patients are observed regarding atrial fibrillation postsurgical. The difference between the group of patients with and without nux vomica is recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients before elective Heart valve - or aortocoronary by pass surgery with heart-lung-machine.

Exclusion Criteria:

* Pregnant patients
* Patients with preoperative atrial fibrillation and/or hyperthyreosis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Frequency of atrial fibrillation after heart surgery with heart lung machine | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frass, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept Surgery, Med Univ Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No